CLINICAL TRIAL: NCT00598845
Title: Prospective Study of Endometrial Cancer Treatment in Relation to Molecular Markers in Curettage Specimens.
Brief Title: Molecular Markers in Treatment in Endometrial Cancer
Acronym: MoMaTEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Helse-Bergen HF (Other); Norwegian Cancer Society (Other)
Responsible Party: Principal Investigator, Helga B Salvesen, Professor, MD, PhD, University of Bergen
Other Study IDs: NSD 15501; NSD 15501; REK 96/1478-2; Helse Vest 911351
Record Dates: First submitted 2007-12-26; First posted 2008-01-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Endometrial Neoplasms; Neoplasm Metastasis
Keywords: Endometrial cancer; Molecular markers; Lymph node metastasis; Prospective study; Prognosis; Cancer of Endometrium; Tumor Markers, Biological
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor specimens from endometrial carcinoma, from curettage and hysterectomy specimens, formalin-fixed and paraffin-embedded and fresh frozen, stored at minus 80 °C, corresponding blood samples with normal DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive numbers: Patients with endometrial cancer
  Interventions: Procedure: Tumor biopsy study

INTERVENTIONS:
Procedure: Tumor biopsy study — Tumor specimens from endometrial cancer patients, collected preoperatively and during primary hysterectomy, are investigated.

SUMMARY:
The purpose of this prospective multicenter trial is to investigate the value of molecular markers in endometrial cancer for predicting lymph node metastasis and prognosis in relation to treatment.

DETAILED DESCRIPTION:
This is a prospective multicenter study to investigate the predictive value of molecular markers in endometrial cancer for lymph node metastasis, prognosis and treatment. For the previously studied tumor markers p53, p16, ER, PR and HER2neu, we want to investigate the expression in curettage material in relation to lymph node metastasis and prognosis among endometrial carcinoma patients. We also want to investigate the distribution of genetic alterations in fresh frozen tumor tissue in order to design prospective randomized treatment trials of metastatic endometrial cancer based on molecular profile. There will be a special emphasis on disturbances in the pathways influenced by new targeted therapy, such as inhibitors of Her2/NEU, EGFR, receptor tyrosine kinase, mTOR, PTEN and hormone receptor pathways.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometrial carcinoma
* Available endometrial biopsy
* Informed consent

Exclusion Criteria:

* No informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with endometrial carcinoma that undergo an endometrial biopsy before treatment with hysterectomy with bilateral salpingoophorectomy with or without pelvic lymph node staging.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-04; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Presence of lymph node metastases | At primary treatment

SECONDARY OUTCOMES:
Recurrent disease, death from disease | 5 years after primary treatment

CONTACTS AND LOCATIONS:
Overall Officials: Helga B. Salvesen, Prof., MD, PhD, Principal Investigator — University of Bergen
Locations (9):
- Gynecological Oncology, UZ Gasthuisberg, Leuven, Belgium
- Norway (7):
  - Department of Gynecology, Ålesund Hospital, Ålesund
  - Sentralsykehuset i Førde, Førde
  - Helse-Fonna, Haugesund Sjukehus, Haugesund
  - Kvinneklinikken, Akershus Universitetssykehus, Lørenskog
  - Kvinnesenteret, Ullevål Universitetssykehus, Oslo
  - Department of Gynecology, St Olav's Hospital, Trondheim
  - Sykehuset Vestfold HF, Tønsberg
- Senter for Surgical Gynecologic Oncology, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Engelsen IB, Stefansson I, Akslen LA, Salvesen HB. Pathologic expression of p53 or p16 in preoperative curettage specimens identifies high-risk endometrial carcinomas. Am J Obstet Gynecol. 2006 Oct;195(4):979-86. doi: 10.1016/j.ajog.2006.02.045. Epub 2006 May 3. PMID 16677592
- [Background] Stefansson IM, Salvesen HB, Akslen LA. Vascular proliferation is important for clinical progress of endometrial cancer. Cancer Res. 2006 Mar 15;66(6):3303-9. doi: 10.1158/0008-5472.CAN-05-1163. PMID 16540684
- [Background] Bachmann IM, Halvorsen OJ, Collett K, Stefansson IM, Straume O, Haukaas SA, Salvesen HB, Otte AP, Akslen LA. EZH2 expression is associated with high proliferation rate and aggressive tumor subgroups in cutaneous melanoma and cancers of the endometrium, prostate, and breast. J Clin Oncol. 2006 Jan 10;24(2):268-73. doi: 10.1200/JCO.2005.01.5180. Epub 2005 Dec 5. PMID 16330673
- [Background] Stefansson IM, Salvesen HB, Akslen LA. Prognostic impact of alterations in P-cadherin expression and related cell adhesion markers in endometrial cancer. J Clin Oncol. 2004 Apr 1;22(7):1242-52. doi: 10.1200/JCO.2004.09.034. PMID 15051772
- [Background] Straume O, Chappuis PO, Salvesen HB, Halvorsen OJ, Haukaas SA, Goffin JR, Begin LR, Foulkes WD, Akslen LA. Prognostic importance of glomeruloid microvascular proliferation indicates an aggressive angiogenic phenotype in human cancers. Cancer Res. 2002 Dec 1;62(23):6808-11. PMID 12460889
- [Background] Salvesen HB, Iversen OE, Akslen LA. Prognostic significance of angiogenesis and Ki-67, p53, and p21 expression: a population-based endometrial carcinoma study. J Clin Oncol. 1999 May;17(5):1382-90. doi: 10.1200/JCO.1999.17.5.1382. PMID 10334522
- [Background] Wik E, Trovik J, Iversen OE, Engelsen IB, Stefansson IM, Vestrheim LC, Haugland HK, Akslen LA, Salvesen HB. Deoxyribonucleic acid ploidy in endometrial carcinoma: a reproducible and valid prognostic marker in a routine diagnostic setting. Am J Obstet Gynecol. 2009 Dec;201(6):603.e1-7. doi: 10.1016/j.ajog.2009.07.029. Epub 2009 Oct 3. PMID 19800606
- [Background] Salvesen HB, Carter SL, Mannelqvist M, Dutt A, Getz G, Stefansson IM, Raeder MB, Sos ML, Engelsen IB, Trovik J, Wik E, Greulich H, Bo TH, Jonassen I, Thomas RK, Zander T, Garraway LA, Oyan AM, Sellers WR, Kalland KH, Meyerson M, Akslen LA, Beroukhim R. Integrated genomic profiling of endometrial carcinoma associates aggressive tumors with indicators of PI3 kinase activation. Proc Natl Acad Sci U S A. 2009 Mar 24;106(12):4834-9. doi: 10.1073/pnas.0806514106. Epub 2009 Mar 4. PMID 19261849
- [Background] Dutt A, Salvesen HB, Chen TH, Ramos AH, Onofrio RC, Hatton C, Nicoletti R, Winckler W, Grewal R, Hanna M, Wyhs N, Ziaugra L, Richter DJ, Trovik J, Engelsen IB, Stefansson IM, Fennell T, Cibulskis K, Zody MC, Akslen LA, Gabriel S, Wong KK, Sellers WR, Meyerson M, Greulich H. Drug-sensitive FGFR2 mutations in endometrial carcinoma. Proc Natl Acad Sci U S A. 2008 Jun 24;105(25):8713-7. doi: 10.1073/pnas.0803379105. Epub 2008 Jun 13. PMID 18552176
- [Derived] Trovik J, Wik E, Werner HM, Krakstad C, Helland H, Vandenput I, Njolstad TS, Stefansson IM, Marcickiewicz J, Tingulstad S, Staff AC; MoMaTEC study group; Amant F, Akslen LA, Salvesen HB. Hormone receptor loss in endometrial carcinoma curettage predicts lymph node metastasis and poor outcome in prospective multicentre trial. Eur J Cancer. 2013 Nov;49(16):3431-41. doi: 10.1016/j.ejca.2013.06.016. Epub 2013 Aug 8. PMID 23932335
- See also: Nordic Society of Gynecologic Oncology — http://www.nsgo.org/